CLINICAL TRIAL: NCT06030609
Title: The Comparison Between Ringer Lactate Solution and Normal Saline With Dextrose Water in the First Week Post-Operative Period of Deceased Donor and Living Donor Kidney Transplantation
Brief Title: The Comparison Between Ringer Lactate Solution and Normal Saline With Dextrose Water in Post-Operative Period of Kidney Transplantation
Acronym: RINNOR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Suwasin Udomkarnjananun, Assistant Professor, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUKT-FLUID
Record Dates: First submitted 2023-09-01; First posted 2023-09-11 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Electrolyte Imbalance; Kidney Transplant; Complications
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ringer lactate arm (Experimental): The patient will receive RLS as a replacement fluid for urine output (mL per mL) until the patient have sufficient oral intake and fluid can be removed.
  Interventions: Drug: Ringer's Lactate Crystalloid Solutions
- Normal saline arm with dextrose water (Active Comparator): The patient will receive NSS with D5W as a replacement fluid for urine output (mL per mL) until the patient have sufficient oral intake and fluid can be removed.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ringer's Lactate Crystalloid Solutions — The patient will receive RLS as a replacement fluid for urine output (mL per mL) until the patient have sufficient oral intake and fluid can be removed.
  Arms: Ringer lactate arm
Drug: Normal saline — The patient will receive NSS with D5W as a replacement fluid for urine output (mL per mL) until the patient have sufficient oral intake and fluid can be removed.
  Other Names: NSS + D5W
  Arms: Normal saline arm with dextrose water

SUMMARY:
This is a randomized controlled pragmatic clinical trial. We aim to evaluate the effect of Ringer lactate solution (RLS) and normal saline solution (NSS) with dextrose water (D5W) on the electrolyte abnormality of kidney transplant recipients (KTR) during the first post-operative week. The problem with using NSS with or without D5W as a standard replacement fluid is the hyperchloremic metabolic acidosis which might compromise the kidney allograft function. A total 60 KTR will be enrolled and randomized to receive either RLS or NSS with D5W. The primary outcome is serum bicarbonate level at day 5 after transplantation. Secondary outcomes include the serum potassium, serum sodium, serum chloride, cytokine panel, and the incidence of delayed graft function.

ELIGIBILITY:
Inclusion Criteria:

* A kidney transplant recipient who receives transplant at King Chulalongkorn Memorial Hospital.
* Age >=18 years
* Both deceased donor and living donor kidney transplantation will be included

Exclusion Criteria:

* multiorgan transplantation
* Known allergy to RLS or NSS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Serum bicarbonate level | Day 5 after transplantation

SECONDARY OUTCOMES:
Serum potassium level | Day 5 after transplantation
Serum chloride level | Day 5 after transplantation
Immune function marker | Day 5 after transplantation
  TNF-alpha

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Nephrology, Faculty of Medicine, King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided